CLINICAL TRIAL: NCT00034970
Title: Mindfulness-Based Art Therapy for Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: R21AT000683-01 (NIH)
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Cancer
Keywords: alternative medicine; art; cancer; combination cancer therapy; creative-expression; group therapy; holistic; human therapy evaluation; meditation; neoplasm /cancer chemotherapy; coping; gender difference; outcomes research; psychological aspect of cancer; psychological stressor; quality of life; racial /ethnic difference; stress management; support; behavioral /social science research; patient oriented research
MeSH Terms: conditions — Neoplasms; Stress, Psychological

INTERVENTIONS:
Behavioral: Mindfulness-based at therapy

SUMMARY:
The purpose of this study is to determine whether cancer patients who receive the mindfulness-based art therapy (MBAT) program demonstrate improvement in health-related quality of life, a reduction in stress-related symptoms, and enhanced coping responses.

DETAILED DESCRIPTION:
Psychosocial interventions, especially supportive-expressive group therapies, have been associated with significant improvements in health status, quality of life and coping behaviors, in patients with cancer. The purpose of the proposed pilot research study is to investigate a newly developed group therapy for cancer patients, MBAT. This proposed, randomized, controlled study follows a successful preliminary investigation of MBAT conducted at Thomas Jefferson University Hospital. MBAT integrates known benefits of art therapy, group therapy, and mindfulness-based stress reduction. Each of these fundamentally different modalities has documented usefulness in the treatment of cancer patients. The multi-modal approach is designed to enhance both the supportive and expressive aspects of the group experience. The study will be done with 96 patients who have a variety of cancer types. Participants will be matched for age and assigned randomly to either the MBAT experimental group or a non-intervention control group. Both groups will continue to receive their usual oncologic/medical care. The MBAT program consists of eight weekly meetings of two and one half-hours in length. At the end of the eight weeks, participants in the control group will be crossed over to the experimental intervention arm for an additional eight weeks. Participants will be assessed pre- and post-intervention on measures of health-related quality of life, psychological distress, and coping, using standardized outcome instruments (SF-36, SCL-90-R and COPE). Our long-term goal is to collect sufficient data to determine the overall efficacy of this promising intervention and to identify which patients are particularly likely to benefit from MBAT.

ELIGIBILITY:
Inclusion:

* Diagnosis of cancer or cancer recurrence within the past 2 years.
* Able to tolerate 8 weekly groups, 2 1/2 hours in length

Exclusion:

* Less than 4 months from original or recurrent diagnosis or beyond 2 years
* Physically unable to attend groups
* Non-stabilized major mental disorder
* Children
* Comprehension of written and spoken English at a level of less than 4th grade.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114
Dates: Start 2002-04; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A. Monti, MD, Principal Investigator — Thomas Jefferson University; Caroline Peterson, MA, Study Director — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital/Kimmel Cancer Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Reibel DK, Greeson JM, Brainard GC, Rosenzweig S. Mindfulness-based stress reduction and health-related quality of life in a heterogeneous patient population. Gen Hosp Psychiatry. 2001 Jul-Aug;23(4):183-92. doi: 10.1016/s0163-8343(01)00149-9. PMID 11543844
- [Background] Speca M, Carlson LE, Goodey E, Angen M. A randomized, wait-list controlled clinical trial: the effect of a mindfulness meditation-based stress reduction program on mood and symptoms of stress in cancer outpatients. Psychosom Med. 2000 Sep-Oct;62(5):613-22. doi: 10.1097/00006842-200009000-00004. PMID 11020090